CLINICAL TRIAL: NCT04504877
Title: Burnout and Distress preventiOn With caNnabidiol in Front-line Health Care workerS deAling (Bonsai Study) wIth COVID-19: a Randomised Controlled Trial
Brief Title: Burnout and Distress preventiOn With caNnabidiol in Front-line Health Care workerS deAling wIth COVID-19
Acronym: BONSAI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jose Alexandre S Crippa, Full Professor - Psychiatry, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BONSAI Study
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Burn Out; Post Traumatic Stress Disorder
MeSH Terms: conditions — COVID-19; Burnout, Psychological; Stress Disorders, Post-Traumatic | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Volunteers, administrative staff, laboratory technicians, doctors who will carry out the assessments by phone, and statisticians will be blind to the treatment group and will not know about the group treatment information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cannabidiol plus general clinical supportive measures (Experimental): The participants will receive CBD 300mg/daily plus general measures (supporting motivational videos, fitness videos). All the participants will perform invasive and non-invasive procedures with the nursing team, the invasive being five blood collections, in their workplaces, to evaluate laboratory parameters, detailed in this project. The non-invasive ones refer to the measurement of height, weight, body temperature, and sleep pattern, as well as five collections of saliva, in a collecting tube, to assess viral load. They will also be monitored through weekly self-assessment scales, applied remotely, electronically (cell phones or computers), with an estimated duration of ten minutes each, which will have their responses recorded in an electronic database by the study coordination team.
  Interventions: Drug: Cannabidiol
- general clinical supportive measures (Other): The participants will receive general measures (supporting motivational videos, fitness videos) alone. All the participants will perform invasive and non-invasive procedures with the nursing team, the invasive being five blood collections, in their workplaces, to evaluate laboratory parameters, detailed in this project. The non-invasive ones refer to the measurement of height, weight, body temperature, and sleep pattern in a collecting tube to assess viral load. Also, they will be monitored through weekly self-assessment scales, applied remotely, electronically (cell phones or computers), with an estimated duration of ten minutes each, which will have their responses recorded in an electronic database by the study coordination team.
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Cannabidiol 300 mg daily for 4 weeks
  Other Names: general clinical supportive measures

SUMMARY:
The objective of this work is to monitor the level of stress and overload of a group of front-line health workers (physicians, nurses and physiotherapists) who will participate in the care of patients with COVID-19 at Hospital das Clínicas in Ribeirão Preto and its Emergency Unit (HCRP), for four weeks, and evaluate the cannabidiol - CBD's effectiveness in reducing stress for those who wish to use it.

DETAILED DESCRIPTION:
The Bonsai study is a two-arm, parallel-group, individually randomized (1:1 allocation ratio), controlled with general measures (supporting motivational videos, fitness videos), participant and investigator unblinded, evaluator by phone will be blinded, single-site superiority trial of oral CBD 300 mg daily for 28 days to prevent burnout and distress in health care workers dealing with SARS-CoV-2 exposure. At 28 days, there is an open-label extension wherein all participants are offered a 28 days course of CBD 300mg daily. The objective of this work is to monitor the level of stress and overload of a group of front-line health workers (physicians, nurses and physiotherapists) who will participate in the care of patients with COVID-19 at Hospital das Clínicas in Ribeirão Preto and its Emergency Unit (HCRP), for four weeks, and evaluate the CBD's effectiveness in reducing stress for those who wish to use it.

This research intends to :

1. Assess the level of stress and emotional overload of front-line health workers (physicians, nurses and physiotherapists) during their performance in the pandemic caused by COVID-19.
2. Assess whether the daily use of CBD 300 mg, for four weeks, reduces the level of stress, during the period of performance of professionals in the care of patients with COVID-19.
3. Assess whether the daily use of CBD 300 mg, for four weeks, will modify inflammatory parameters, such as cytokines, measured from the serum of professionals in the care of patients with COVID-19.
4. Assess whether the daily use of CBD 300 mg, for four weeks, prevents depression, burnout and Acute Stress Disorder and PTSD.
5. Assess the possible adverse effects of using CBD

ELIGIBILITY:
Inclusion Criteria:

1. age between 24 and 60 years old
2. Research participants of both sexes.
3. HCFMRP physicians, nurses and physiotherapists involved in the care of patients who have undergone screening and present at least one symptom, which may be related to infection by COVID-19.
4. Good health conditions and without conditions that characterize them as belonging to the risk groups associated with COVID infection19.
5. Research participants with the potential to become pregnant may be included in the study as long as they are sexually abstinent or using a contraceptive method considered effective.
6. Signature of the Free and Informed Consent Term approved (ICF) by the Research Ethics Committee (CEP) and CONEP.

Exclusion Criteria:

1. Using any medication with potential interaction with CBD or with a history of undesirable reactions prior to the use of this cannabinoid.
2. Physicians, nurses and physiotherapists with occasional contact with patients with COVID-19 and who are not responsible for the continuous monitoring of these patients.
3. Although in the HC-FMRP-USP care allocation policy, professionals who are eventually more susceptible to complications from the new coronavirus will be relocated to not attend patients with COVID19, it will be checked again to exclude patients with chronic diseases: diabetes, hypertension, lung disease like asthma or COPD; hematological diseases, chronic kidney disease and immunodepression.
4. Professionals over 60 years old
5. Female research participants who become pregnant or male participants who have their pregnant partner during the research project

Ages: 24 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
aMBI-HSS: Abbreviated Maslach Burnout Inventory - Human Services Survey | Through study completion, over time during the study period (day 0-28)
  To assess the emotional exhaustion dimension of the burnout syndrome, based on nine items, scored from 0 ("never") to 6 ("every day")

SECONDARY OUTCOMES:
Brief measure for assessing generalized anxiety disorder: The GAD-7 | Through study completion, over time during the study period (day 0-28)
  brief measure for assessing generalized anxiety disorder
PHQ-9: Patient´s Health Questionnaire-9 | Through study completion, over time during the study period (day 0-28)
  Evaluate depressive symptoms o
Change in proinflammatory cytokine concentration | Through study completion, over time during the study period (day 0-28)
  Laboratory parameters, including the change in proinflammatory cytokine concentrations
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Through study completion, over time during the study period (day 0-28)
  Occurrence of side effects
Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Through study completion, over time during the study period (day 0-28)
  It is a self-report measure widely used to assess PTSD symptoms, according to the DSM-5 criteria. The reduced version of this instrument will be used (8 items)

CONTACTS AND LOCATIONS:
Overall Officials: Jose A. Crippa, MD; PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately the following publication. No end date
Access Criteria: Researchers who provide a methodologically sound proposal. Depending on the level of the proposed use of data, approval by an independent review committee will be required for the identified purpose.

REFERENCES:
- [Derived] Crippa JAS, Zuardi AW, Guimaraes FS, Campos AC, de Lima Osorio F, Loureiro SR, Dos Santos RG, Souza JDS, Ushirohira JM, Pacheco JC, Ferreira RR, Mancini Costa KC, Scomparin DS, Scarante FF, Pires-Dos-Santos I, Mechoulam R, Kapczinski F, Fonseca BAL, Esposito DLA, Pereira-Lima K, Sen S, Andraus MH, Hallak JEC; Burnout and Distress Prevention With Cannabidiol in Front-line Health Care Workers Dealing With COVID-19 (BONSAI) Trial Investigators. Efficacy and Safety of Cannabidiol Plus Standard Care vs Standard Care Alone for the Treatment of Emotional Exhaustion and Burnout Among Frontline Health Care Workers During the COVID-19 Pandemic: A Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2120603. doi: 10.1001/jamanetworkopen.2021.20603. PMID 34387679